CLINICAL TRIAL: NCT07180914
Title: A Real-world Study on the Compliance of OFS-assisted Endocrine Therapy for HR+ Premenopausal Breast Cancer
Brief Title: A Real-world Study on the Compliance of OFS-assisted Endocrine Therapy for Hormone Receptor-positive(HR+) Premenopausal Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Beijing Health Promotion Association (Unknown)
Responsible Party: Principal Investigator, Yu Yang, MD, Zhejiang Cancer Hospital
Other Study IDs: IRB-2025-977
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Females
Keywords: OFS; Hormone receptor positive; Early-stage breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early-stage HR-positive premenopausal breast cancer patients receiving OFS treatment.

SUMMARY:
The goal of this observational study is to observe the long-term prognosis of patients with early HR-positive premenopausal breast cancer. The study also aims to understand the compliance with and reasons for discontinuing adjuvant OFS endocrine therapy under different combination regimens.

The main questions it aims to answer are:

1. What are the rates of compliance with and reasons for discontinuation of adjuvant OFS endocrine therapy?
2. What is the impact of OFS treatment duration on patient prognosis?

Participants, who are already receiving OFS treatment as part of their regular medical care, will have their demographic data, treatment status, clinical outcomes, and adverse events collected over time.

DETAILED DESCRIPTION:
This real-world non-interventional prospective study aims to explore the compliance and reasons for discontinuation of adjuvant OFS endocrine therapy in early HR-positive premenopausal breast cancer patients under different combination regimens of adjuvant endocrine drugs, as well as to observe the impact of the duration of OFS treatment on prognosis. This study adopts a multi-center, prospective, non-interventional design to collect approximately 300 cases of early HR-positive premenopausal breast cancer patients who received OFS treatment. After obtaining informed consent, the demographic data, breast cancer diagnosis information, comorbidities, past medical history, treatment status, clinical outcomes, and adverse events of the patients were collected. The patients were administered medication in accordance with the standard clinical drug protocols and completed follow-up according to the follow-up plan.

ELIGIBILITY:
Inclusion Criteria:

1. Female breast cancer patients who were premenopausal at the time of surgery.
2. Newly diagnosed patients with invasive breast cancer, tumor node metastasis(TNM) stage I-III.
3. HR-positive (defined as ER ≥ 10% and/or progesterone receptor(PR) ≥ 10%).
4. Patients who have undergone radical mastectomy and are planning to receive OFS treatment.
5. Have received (neo)adjuvant chemotherapy and radiotherapy.
6. Eastern Cooperative Oncology Group Performance Status(ECOG PS) score of 0-1.
7. Complete medical records.
8. Willing to accept long-term follow-up.
9. Any adverse events that occurred during adjuvant chemotherapy (if applicable) have recovered or decreased to grade 1 (according to CTCAE v5.0) at the start of OFS treatment.

Exclusion Criteria:

1. Simultaneously participating in another blinded clinical study.
2. Presence of other active malignant tumors or multiple primary cancers.
3. Pregnant or lactating women.
4. Other conditions that the investigator deems unsuitable for inclusion in the study.
5. Planning to use systemic therapies not described in the study cohort during the endocrine therapy phase (such as, but not limited to, chemotherapy, Antibody-Drug Conjugates(ADCs), or immunotherapy).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Female breast cancer patients who were premenopausal at the time of surgery.
  2. Newly diagnosed patients with invasive breast cancer, TNM stage I-III.
  3. HR-positive (defined as ER ≥ 10% and/or PR ≥ 10%).
  4. Patients who have undergone radical mastectomy and are planning to receive OFS treatment.
  5. Have received (neo)adjuvant chemotherapy and radiotherapy.
  6. ECOG PS score of 0-1.
  7. Complete medical records.
  8. Willing to accept long-term follow-up.
  9. Any adverse events that occurred during adjuvant chemotherapy (if applicable) have recovered or decreased to grade 1 (according to CTCAE v5.0) at the start of OFS treatment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to different Ovarian Function Suppression (OFS) combination regimens and reasons for discontinuation. | Follow-up will be conducted every 3 months during the period from baseline to 2 years of endocrine therapy.
  The proportion of patients who discontinue OFS within 2 years.

SECONDARY OUTCOMES:
Effect of OFS Treatment Duration on Prognosis. | 3-year iDFS rate for OFS treatment duration ≥2 years and <2 years
  To observe the effect of OFS treatment duration on prognosis.
3-year iDFS for Different OFS Combination Regimens. | 3 years.
  3-year iDFS for different OFS combination therapy regimens.
Safety of different combination regimens | During the follow-up period, which is every 3 months within the first 2 years, and every 6 months from year 2 to year 3
  The collection and analysis of various adverse events and serious adverse events that occur during different treatment processes.
3-year iDFS of different subgroups | 3 years
  The 3-year invasive disease-free survival (iDFS) for different patient subgroups.